CLINICAL TRIAL: NCT05355753
Title: A Phase 1/2 Open-Label, Multicenter Study to Characterize the Safety and Tolerability of CFT8634 in Subjects With Locally Advanced or Metastatic SMARCB1-Perturbed Cancers, Including Synovial Sarcoma and SMARCB1-Null Tumors
Brief Title: A Study to Assess the Safety and Tolerability of CFT8634 in Locally Advanced or Metastatic SMARCB1-Perturbed Cancers, Including Synovial Sarcoma and SMARCB1-Null Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: High levels of BRD9 degradation did not result in sufficient efficacy in heavily pre-treated synovial sarcoma and SMARCB1-null solid tumor patients treated with CFT8634 as a single agent.
Sponsor: C4 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CFT8634-1101
Record Dates: First submitted 2022-04-23; First posted 2022-05-02 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Synovial Sarcoma; Soft Tissue Sarcoma
Keywords: Synovial Sarcoma; SMARB1-Null Tumors; CFT8634; Soft Tissue Sarcoma; Myoepithelial Carcinoma; Extraskeletal Myxoid Chondrosarcoma; Renal Medullary Carcinoma; Chordoma; Epithelioid Sarcoma
MeSH Terms: conditions — Sarcoma, Synovial; Sarcoma; Chondrosarcoma, Extraskeletal Myxoid; Chordoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation Phase 1/Part1: CFT8634 (Experimental): Up to approximately 40 subjects ≥18 years of age or between ≥16 and <18 years of age and weighing ≥50 kg with locally advanced or metastatic SMARCB1-perturbed cancers, including synovial sarcoma and SMARCB1-null tumors, having received ≥ 1 prior anticancer therapy
  Interventions: Drug: CFT8634
- Dose Escalation Phase 1/Part 2: CFT8634 (Experimental): Up to approximately 6-12 subjects ≥12 and <16 years of age and weighing ≥40 kg or ≥16 and <18 years of age and weighing ≥40 kg and <50 kg with locally advanced or metastatic SMARCB1-perturbed cancers, including synovial sarcoma and SMARCB1-null tumors
  Interventions: Drug: CFT8634
- Phase 2 - Arm A: CFT8634 (Experimental): Approximately 30 subjects with locally advanced or metastatic synovial sarcoma at the recommended phase 2 dose (RP2D) having received 1-2 prior anticancer therapies
  Interventions: Drug: CFT8634
- Phase 2 - Arm B: CFT8634 (Experimental): Approximately 20 subjects with locally advanced or metastatic SMARCB1-null tumors at the RP2D having received ≥1 prior anticancer therapy
  Interventions: Drug: CFT8634

INTERVENTIONS:
Drug: CFT8634 — Oral dose of CFT8634

SUMMARY:
This is an open-label, non-randomized, first-in-human Phase 1/2 study designed to evaluate the safety and tolerability of CFT8634 in subjects with synovial sarcoma and SMARCB1-null tumors who: have received prior systemic therapy; have relapsed/refractory tumors; have unresectable or metastatic disease; and are not candidates for available therapies known to confer clinical benefit. The study will characterize the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary antitumor activity of CFT8634.

DETAILED DESCRIPTION:
The study was intended to be Phase 1/2 trial but did not advance to Phase 2.

ELIGIBILITY:
Inclusion Criteria:

1. Subject (and legal guardian where applicable) is (are) willing and able to provide signed informed consent (or assent, where applicable) and can follow protocol requirements
2. Subject has histologically or cytologically confirmed synovial sarcoma or SMARCB1-null sold tumor that is relapsed/refractory, and unresectable or metastatic; the subject must not be a candidate for available therapies that are known to confer clinical benefit

   a. Phase 1: subject must have received ≥1 prior line of systemic anticancer therapy considered to be Standard of Care per the Investigator's judgment, in the metastatic or unresectable setting b. Phase 2: i. Arm A: subject must have received only 1-2 prior lines of systemic anticancer therapy considered to be Standard of Care per the Investigator's judgment, in the metastatic or unresectable setting ii. Arm B: subject must have received ≥1 prior line of systemic anticancer therapy considered to be Standard of Care per the Investigator's judgment, in the metastatic or unresectable setting
3. Subject must be:

   * ≥18 years of age (no minimum weight),
   * ≥16 and <18 years old and weighs ≥50 kg,
   * ≥12 and <16 years of age and weighs ≥40kg,
   * or ≥16 and <18 years of age and weighs ≥40kg and <50kg
4. Subject must be able to safely swallow capsules
5. Subject must have measurable disease as defined by RECIST v1.1
6. Subject must have Eastern Cooperative Oncology Group performance status ≤2 or Lansky performance scale (LK scale) ≥ 60
7. Subject must have adequate organ function, defined as:

   1. Bone marrow function: absolute neutrophil count ≥1.0 x 109/L independent of growth factor support for ≤7 days prior to first dose of study drug for granulocyte colony-stimulating factor and ≤14 days prior to first dose of study drug for peg-filgrastim; hemoglobin ≥8 g/dL independent of transfusion support for ≤7 days prior to first dose of study drug; platelet count ≥75 x 109 /L independent of transfusion support for ≤3 days prior to first dose of study drug
   2. Coagulation: Prothrombin time (PT)/international normalized ratio (INR) <1.5x the upper limit of normal (ULN) and activated partial thromboplastin time (aPTT) <1.5x ULN (unless the subject is receiving anticoagulant therapy and INR and partial PT/aPTT are within therapeutic range of intended use of anticoagulants)
   3. Liver function: total bilirubin ≤1.5x ULN (≤3.0x ULN for subjects with Gilbert's syndrome), aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0x ULN; except for subjects who have tumor infiltration of the liver, where ALT and AST ≤5x ULN
   4. Renal function: must have a creatinine clearance ≥60 mL/min (via Cockcroft-Gault equation, institutional standard, or measured)
   5. Cardiac function: baseline corrected QT interval using Fredericia's formula ≤470 ms (adolescents 12-17 years of age: ≤450 ms) and a left ventricular ejection fraction ≥50% evaluated via echocardiogram or multi-gated acquisition (MUGA) scan
8. Availability of archival tumor tissue sample or newly obtained core/excisional biopsy of a tumor not previously irradiated
9. A female subject may be eligible to participate if she is not pregnant or planning a pregnancy, not breastfeeding, and following protocol mediated guidance to avoid pregnancy
10. A male subject must have had a prior vasectomy and agree to use a condom during the treatment period and for at least 90 days after the last dose of study treatment
11. A male subject must refrain from donating sperm while taking CFT8634 and for 90 days post-last dose
12. A female subject must refrain from donating ova while taking CFT8634 and for 180 days after discontinuation
13. All subjects must refrain from donating blood and blood products while receiving study drug and for 30 days post-last dose

Exclusion Criteria:

1. Subject has had major surgery within 21 days prior to the planned first dose of CFT8634

   a. Minor surgery (eg, minor biopsy of extracranial site, central venous catheter placement, shunt revision) is permitted within 21 days prior to first dose of CFT8634
2. Subject has received standard of care or investigational systemic anti-neoplastic therapy within 14 days or 5 half-lives, whichever is shorter, prior to the planned first dose of CFT8634
3. Subject has received radiation therapy within 14 days prior to the planned first dose of CFT8634
4. Prior treatment with BRD9 degrader
5. Subject has central nervous system (CNS) involvement (primary tumor or metastatic disease), except in the following circumstances:

   1. Subjects with previously treated brain metastases may be permitted to participate provided they are stable (without evidence of progression by imaging 14 days prior to the first dose of study drug and any neurologic symptoms have stabilized), have no evidence of new or enlarging brain metastases, and if they are taking corticosteroids, they are on stable or tapering doses for at least 7 days prior to first dose of study drug. Antiseizure therapy is permitted provided the medication is not otherwise excluded and seizures have been controlled for at least 28 days since the last antiseizure medication adjustment
   2. Subjects with asymptomatic brain metastases found on Screening magnetic resonance imaging (MRI) may be permitted to be entered into the study without prior radiation therapy to the brain if they do not require immediate surgical or radiation therapy in the opinion of the treating investigator and in the opinion of a radiation therapy or neurosurgical consultant
6. Subject has any evidence of a CNS bleed including intra-tumoral hemorrhage
7. Subject has known bleeding diathesis
8. Subject has impaired cardiac function or clinically significant cardiac disease (i.e. uncontrolled heart disease/hypertension, clinically significant arrythmias, unstable angina/myocardia infarction/stroke within 180 days prior to screening)
9. Subject with presence of inflammatory vascular disease or microangiopathy (eg, thrombotic microangiopathies, hemolytic uremic syndrome [HUS], atypical HUS)
10. Subject with known malignancy, other than study indication, that is progressing or has required treatment within the past 3 years

    a. Subject with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (i.e. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
11. Subject has received live, attenuated vaccine within 28 days prior to first dose administration
12. Subject with known history of human immunodeficiency virus (HIV) infection
13. Subject had a venous thrombosis within 14 days prior to first dose of study drug
14. Subject with gastrointestinal absorption issues (e.g., malabsorption syndrome or other illness that could affect oral absorption).
15. Concurrent administration of strong cytochrome P450 (CYP) 3A4 inhibitors and inducers, and multidrug resistance mutation 1 (MDR1) inhibitors.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of AEs and serious adverse events (SAEs) | From screening until at least 30 days after completion of study treatment
  Phase 1 and Phase 2
Number of subjects with changes between baseline and post-baseline safety assessments based on safety laboratory results graded by CTCAE v5.0 | From screening until at least 30 days after completion of study treatment
  Phase 1 and Phase 2
Frequency of dose interruptions and dose reductions | From first dose until end of treatment
  Phase 1 and Phase 2
Incidence of dose limiting toxicities (DLTs) | From first dose until 28 days after first dose
  Phase 1 only
Overall Response Rate (ORR) | Up to approximately 24 months
  Phase 2 only according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
Plasma concentration of CFT8634 to characterize the pharmacokinetics (PK) parameters of CFT8634 | At multiple time points up to approximately 24 weeks
  Plasma concentration of CFT8634 at the scheduled timepoints
Asses dose proportionality assessment | At multiple time points up to approximately 24 weeks
  Dose proportionately assessment at the scheduled timepoints
Assess the pharmacodynamics by percent reduction from baseline of target protein | At multiple time points up to approximately 24 weeks
  Tumor BRD9 degradation at scheduled timepoints
ORR | Up to approximately 24 months
  Phase 1 only according to RECIST v1.1 criteria
Duration of Response (DOR) | Up to approximately 24 months
  DOR defined as time from first assessment of PR or CR to follow-on first assessment of progressive disease (PD)
Progression Free Survival (PFS) | Up to approximately 24 months
  PFS defined as the time from first treatment received until PD is assessed
Overall Survival (OS) | Up to approximately 48 months
  OS is defined as the time from first dose of study treatment to the date of death, irrespective of the cause of death. (Phase 2 only)
Time to next treatment | Up to approximately 8 months
  Interval from the date of initiation of a treatment to the date of commencement of the next line of therapy

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - City of Hope, Duarte, California
  - Sarcoma Oncology Research Center, Santa Monica, California
  - University of Colorado - Aurora Cancer Center, Aurora, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - David H. Koch Center for Cancer Care at Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No